CLINICAL TRIAL: NCT01980030
Title: Using ROMIPLOSTINE for Persistent Thrombocytopenia With Transfusion-dependent Patients Who Received Allogeneic Hematopoietic Stem Cell
Acronym: AGRAH003
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P110204
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Persistent Thrombocytopenia Following Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
MeSH Terms: interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Romiplostim (Experimental): Weekly Romiplostim for 12 weeks with intra-patient weekly dose escalation from 1µg/Kg to a maximum dose of 10 µg/Kg with a dose reduction schema in case of platelet overshoot
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim

SUMMARY:
This is a Phase I/II multicenter study which aims to assess the toxicity profile of Romiplostim in patients with transfusion-dependent thrombocytopenia after allogeneic HSCT.

A total of 24 patients with transfusion-dependent thrombocytopenia after allogeneic HSCT will be included.

The main endpoint is the incidence and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥ 18 years, willing and able to sign informed consent
* Patients could have been transplanted for hematological disorder (malignant or non-malignant) excepted myelodysplastic syndromes patients and had received either a myeloablative or a reduced intensity conditioning. All sources of allogeneic stem cells are allowed.
* Prolonged (> 2 months) transfusion-dependent thrombocytopenia
* Screenings mean platelet count≤ 20 x giga/L or screenings mean platelet count ≤ 50 x giga/L with a history of bleeding.
* (ECOG) performance status of 0-2
* Adequate liver function
* Serum creatinine ≤ 176.8 μmol/L
* Bone marrow aspirate with cytogenetics within 6 days of the first dose of romiplostim
* Written informed consent

Exclusion Criteria:

* Relapse/progression of hematological malignancy (marrow examination required)
* Non-controlled acute and/or chronic graft versus host disease (GvHD)
* Active or uncontrolled infections
* Cardiac pathology - Thrombosis
* Pregnancy or breast feeding
* Received interleukin-11 (IL-11) within 4 weeks of screening or previously received any thrombopoietic growth factor
* Patients on anticoagulant therapy
* Receipt or planned receipt of Pegylated Granulocyte Colony Stimulating Factor (PEG-G-CSF), or Granulocyte macrophage-colony stimulating factor (GM-CSF) within 4 weeks of the first dose of investigational product
* Subject not using adequate contraceptive precautions, in the judgment of the investigator
* Sensitivity to any Escherichia coli-derived product
* Inability to comply with study procedures.
* Subject currently is enrolled in or has not yet completed 30 days since ending other investigational device or drug study
* No medical insurance in the French Health system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Adverse events | 12 months
  Incidence and severity of all adverse events

SECONDARY OUTCOMES:
Dose of Romiplostim | 12 months
  Dose of Romiplostim required to reach a platelet count above 50 x 109/L in absence of platelet transfusion
Durable platelet response after transplant: | 12 months
  platelet count above 50 x 109/L on 8 consecutive weeks independent of platelet transfusions
Relapse rate | 12 months
Graft versus host disease (GVHD) | 12 months
Non relapse mortality rate | 12 months
number of platelet transfusions | 12 months
Overall number of bleeding events | 12 months
platelet hematological improvements | 12 months
  Incidence and duration of platelet hematological improvements above 20 x 109/L and above 50 x 109/L , respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis hospital, Paris, Île-de-France Region, France